CLINICAL TRIAL: NCT05089591
Title: Efficacy of Intense Pulsed Light Treatment in Patients With Meibomian Gland Dysfunction
Brief Title: Intense Pulsed Light in Meibomian Gland Dysfunction
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Prim. Prof. Dr. Oliver Findl, MBA (Other)
Responsible Party: Sponsor-Investigator, Prim. Prof. Dr. Oliver Findl, MBA, Prim. Univ. Prof. Dr. Oliver Findl, MBA, Vienna Institute for Research in Ocular Surgery
Organization: Vienna Institute for Research in Ocular Surgery (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IPL
Record Dates: First submitted 2021-10-20; First posted 2021-10-22 (Actual); Last update posted 2021-10-22 (Actual); Status verified 2021-10

CONDITIONS: Meibomian Gland Dysfunction
MeSH Terms: conditions — Meibomian Gland Dysfunction | interventions — Intense Pulsed Light Therapy

STUDY DESIGN:
Intervention Model Description: Bilateral comparison
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Study eyes (Active Comparator): Study eye receives the standard energy dose as recommended by the manufacturer (between 8 and 12J/cm2, in accordance with the manufacturer's recommendations).
  Interventions: Device: Intense Pulsed Light therapy
- Control eyes (Sham Comparator): The control eye is treated using low energy dose energy (1J/ cm2) as sham treatment, ensuring blinding of the respective patient.
  Interventions: Device: Sham Treatment

INTERVENTIONS:
Device: Intense Pulsed Light therapy — The LacryStim System is a CE marked device for treatment of meibomian gland dysfunction. It stimulates and reactivates meibomian glands and improves the related dry eye condition. Intense pulsed light is emitted with a light spectrum from 610nm to 1200nm. Each treatment consists of short individual pulses lasting for 4ms separated by a 26ms lasting interval to hinder tissue temperature increase, thermal damage to the skin and inflammatory reaction. During this phase 8 to 12 J / cm2 are delivered. Selection of total energy levels depends on the skin type (Fitzpatrick Skin Types) as recommended by the manufacturer.
  Arms: Study eyes
Device: Sham Treatment — The fellow eye serves as the control eye. Study eye receives the standard energy dose as recommended by the manufacturer (between 8 and 12J/cm2, in accordance with the manufacturer's recommendations). The control eye is treated using low energy dose energy (1J/ cm2) as sham treatment, ensuring blinding of the respective patient.
  Arms: Control eyes

SUMMARY:
Meibomian gland dysfunction (MGD) is a major cause of dry eye disease (DED). Up to 86% of patients suffering from DED also show signs of MGD. Traditional treatment of MGD is based on eye lid hygiene and massage in combination with intensive usage of lubricants.

Recently, a novel technology the intense pulsed light (IPL) therapy was introduced, which shows promising results in patients with meibomian gland dysfunction. Originating from field of dermatology, subjecting improvement of dry eye symptoms was recognized after the treatment of facial rosacea using IPL. Different hypotheses exist how IPL treatment might improve the situation in the dry eye patient. Warming of the eyelid, due to the light application and reduction of bacterial load are two possible mode of actions. Further, the used wavelengths in IPL may be modified that the light is only absorbed by oxygenated haemoglobin, which lead to an obliteration of telangiectasia and reduced inflammation on the lid margin. This principal is applied in the treatment of facial rosacea.

Aim of this study is to investigate the effect of IPL therapy in patients with MGD on dry eye parameters as well as subjective complaints.

ELIGIBILITY:
Inclusion Criteria:

* Age older than 18 years
* Presence of meibomian gland dysfunction at any stage
* Presence of meibomian glands on each lower eyelid's Meibography

Exclusion Criteria:

* Fitzpatrick Skin Type VI
* Usage of eye drops other than lubricants (e.g. antibiotics, steroids, cyclosporin-A)
* Usage of systemic antibiotic therapy
* Any pathology of the ocular surface except dry eye disease (e.g. corneal scarring, cornea ectasia)
* Ocular surgery within prior 3 months
* Ocular injury within prior 3 months
* Ocular herpes of eye or eyelid within prior 3 months
* Active ocular infection
* Active ocular inflammation or history of chronic, recurrent ocular inflammation within prior 3 months
* Eyelid abnormalities that affect lid function
* Ocular surface abnormality that may compromise corneal integrity
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Estimated)
Dates: Start 2021-10-20 (Actual); Primary Completion 2022-10-20 (Estimated); Study Completion 2022-11-01 (Estimated)

PRIMARY OUTCOMES:
Difference Meibum quality score and expressibility between both eyes during the 6-month visit | 6-months visit

SECONDARY OUTCOMES:
Comparison of dry eye related parameters between both eyes (tear film break up time, Oxford Staining) | 6 months
Change of dry eye related parameters during the study period in the study eye (tear film break up time, Oxford Staining) | 6 months
Change of Ocular Surface Disease Index (OSDI) score during the study period | 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- Vienna Institute for Research in Ocular Surgery, Vienna, Austria

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Schlatter A, Palkovits S, Amir-Asgari S, Ruiss M, Zeilinger J, Rotter A, Schmidl D, Findl O. Safety and efficacy of a novel intense pulsed light system in patients with meibomian gland dysfunction: a randomized, double-masked, intra-individual controlled study. Int Ophthalmol. 2025 Jun 16;45(1):246. doi: 10.1007/s10792-025-03622-2. PMID 40524073